CLINICAL TRIAL: NCT02192437
Title: Dietary Methionine and Cysteine Restriction in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Orentreich Foundation for the Advancement of Science, Inc. (Other)
Responsible Party: Principal Investigator, John P. Richie, Professor of Public Health Sciences & Pharmacology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 03-13-2014
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Healthy
Keywords: methionine; cysteine; sulfur amino acid restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methionine restricted diet (Experimental): Intervention will be a Sulfur amino acid restricted diet (methionine). Control diet for 4 weeks followed by a washout for 3-4 weeks, then a methionine restricted diet (70%) for 4 weeks, followed by 3-4 weeks washout period and then a methionine restricted diet (90%) for 4 weeks.
  Interventions: Other: Sulfur amino acid restricted diet
- Methionine and cysteine restricted diet (Experimental): Intervention will be a Sulfur amino acid restricted diet (methionine and cysteine). Control diet for 4 weeks followed by a washout for 3-4 weeks then a methionine and cysteine restricted diet (50%) followed by 3-4 weeks washout period and then a methionine and cysteine restricted diet (65%) for 4 weeks.
  Interventions: Other: Sulfur amino acid restricted diet

INTERVENTIONS:
Other: Sulfur amino acid restricted diet — Methionine restricted diet: 70% or 90% restriction Methionine and cysteine restricted diet: 50% or 65% restriction

SUMMARY:
Studies in laboratory models indicate that dietary methionine restriction (MR) enhances longevity and produces short- and long-term metabolic changes that are consistent with a healthy lifespan. The present study was designed to establish levels of dietary methionine or methionine and cysteine that induce physiological changes in healthy adults like those observed in rodent studies .

DETAILED DESCRIPTION:
In this controlled feeding study, subjects will be randomized to one of two experimental. Group A (N=10): will start with control diet (31 mg/kg/day Met; 31 mg/kg/day Cys) for 4 weeks followed by a washout for 3-4 weeks, then a 70% MR diet (9.3 mg/kg/day Met; 40.3 mg/kg/day SAA) for 4 weeks, followed by 3-4 weeks washout period and then a 90% MR diet (3.1 mg/kg/day Met; 34.1 mg/kg/day SAA) for 4 weeks. Group B (N=10): will start with control diet (31 mg/kg/day Met; 31 mg/kg/day Cys) for 4 weeks followed by a washout for 3-4 weeks then a 50% methionine and cysteine restricted (M/CR) diet (15.5 mg/kg/day Met; 15.5 mg/kg/day Cys; 31 mg/kg/day SAA), followed by 3-4 weeks washout period and then a 65% M/CR diet (10.8 mg/kg/day Met; 10.8 mg/kg/day Cys; 21.6 mg/kg/day SAA) for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy English speaking male and female volunteers
* May or may not be students
* Age range 24-65 years
* Subjects will need to be of normal weight or moderately overweight (BMI 18.5-35 kg/m2)
* Subjects will be non-smokers

Exclusion Criteria:

* No use of medications known to impact the biomarkers of interest
* Pregnancy and lactating women
* Persons with documented diabetes
* No use of high dose dietary antioxidant supplements or fish oil/flax seed oil for n-acetylcysteine for at least 1 month prior to the study
* Use of tobacco products over the past 6 months
* Unstable weight
* Individuals with allergies to eggs, wheat, nuts, soy and latex
* Individuals with phenylketonuria (PKU)

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07-16 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Body weight, plasma sulfur amino acids | Baseline, four weeks

SECONDARY OUTCOMES:
Biomarkers of oxidative stress, blood lipids | Baseline, four weeks

OTHER OUTCOMES:
Plasma IGF1, insulin | Baseline, four weeks

CONTACTS AND LOCATIONS:
Overall Officials: John P Richie, PhD, Principal Investigator — Penn State University; Sailendra Nichenametla, Ph.D., Principal Investigator — Orentreich Foundation for the Advancement of Science, Inc.
Locations (1):
- Penn State University, State College, Pennsylvania, United States